CLINICAL TRIAL: NCT07309211
Title: A Multi-centre, Retrospective Study Assessing Durvalumab as Consolidation Treatment for Patients With Limited-stage Small Cell Lung Cancer (LS-SCLC) Following by Sequential Chemoradiotherapy (sCRT)
Brief Title: Durvalumab as Consolidation Therapy in Patients With LS-SCLC Following sCRT
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xin Zhao, Chief Physician, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 2025-SR-343.A1
Record Dates: First submitted 2025-12-01; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: SCLC, Limited Stage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
This is a retrospective, multi-centre, single arm study to assess the safety and efficacy of receiving Durvalumab in patients with Small Cell Lung Cancer Limited Stage (LS-SCLC) who have not progressed following sequential chemoradiotherapy (sCRT) in a real-world setting. The study will enroll 25 patients. The primary endpoint of the study is the incidence of Grade 3 or 4 adverse events (AEs) within 6 months of starting Durvalumab (graded by CTCAE v.5.0). The secondary endpoints of the study include real-world progression-free survival (rwPFS, the time from the start of Durvalumab treatment to disease progression or death for any reason, which occurs first), objective response rate (ORR), duration of response (DoR) and disease control rate (DCR).

sCRT is more common in Mid-Eastern Chinese clinical practice. sCRT is also recommended in guideline of Chinese Society of Clinical Oncology (CSCO) Small-cell lung cancer. However, patients treated with sCRT were not included in the ADRIATIC study. So there is lack of data on safety and efficacy of Durvalumab post sCRT. Supplement real-world evidence (RWE) clinical data of sCRT in Chinese patients is needed to enhance the status of Durvalumab as a consolidation therapy for LS-SCLC.

The study will retrospectively collect cases of eligible LS-SCLC patients who received sCRT and have not progressed followed by receiving Durvalumab as consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 at initial diagnosis;
2. Histological or cytological evidence of LS-SCLC (Stage I-III); Stage I-II must be medically inoperable;
3. Received chemotherapy sequential with radiotherapy as first-line treatment and no progression, followed by receiving Durvalumab at least 1 dose as consolidation treatment until progression, unacceptable toxicity or for a maximum of 24 months;
4. Start Durvalumab treatment within 3 months after sCRT;
5. Permitted PCI;
6. WHO PS 0-2 before sCRT.

Exclusion Criteria:

1. ES-SCLC or mixed SCLC and NSCLC histology;
2. Active or prior documented autoimmune or inflammatory disorders or uncontrolled intercurrent illness;
3. Any unresolved toxicity (CTCAE Grade ≥ 2) from prior chemoradiotherapy; 4. Received concurrent chemoradiotherapy for LS-SCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will retrospectively collect cases of eligible LS-SCLC patients who received sCRT and have not progressed followed by receiving Durvalumab as consolidation therapy. The retrospective collection of cases for initiating the administration of Durvalumab spans from December 9, 2019, to April 10, 2025. Retrospective analysis of each case should meet all of the inclusion criteria and exclusion criteria for this study. Under no circumstances can there be exceptions to this rule.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 3 or 4 Adverse Events (AEs) within 6 months of starting Durvalumab [graded by Common Terminology Criteria for Adverse Event (CTCAE) v.5.0] | Within 6 months of starting Durvalumab

SECONDARY OUTCOMES:
Real world PFS (rwPFS) | From date of the first dose of Durvalumab to date of objective disease progression or death, whichever came first, assessed up to 60 months
ORR (Objective response rate from starting with Durvalumab treatment) | Up to 60 months
DoR (Duration of response from starting with Durvalumab treatment) | From the earliest date of first documented evidence of confirmed CR or PR until the earliest date of disease progression or death from any cause, whichever comes first, Up to 60 months
DCR (Disease control rate from staring with Durvalumab treatment) | Up to 60 months

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Cancer Hospital of Shandong First Medical University, Jinan
  - Nanjing Chest Hospital, Nanjing
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing
  - The affiliated hospital of qingdao university, Qingdao